CLINICAL TRIAL: NCT07337863
Title: A Randomized, Double-Blind, Multicenter, Phase II/III Clinical Study Comparing Umbilical Cord-Derived Mesenchymal Stem Cell Secretome Versus Sodium Hyaluronate on Clinical Outcomes, Pain, and Function in Patients With Kellgren-Lawrence Grade 2-3 Knee Osteoarthritis
Brief Title: A Phase II/III Randomized Double-Blind Multicenter Study Comparing UC-MSC-Derived Secretome and Sodium Hyaluronate in Patients With Knee Osteoarthritis
Acronym: SECRET-OA
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universitas Sriwijaya (Other)
Collaborators: PT Bifarma Adiluhung (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCMSC-OA-Phase II/III; PML-BFA-04-2024 (Other Grant/Funding Number: PT Bifarma Adiluhung)
Record Dates: First submitted 2026-01-01; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Knee Osteoarthritis (Knee OA)
Keywords: Knee Osteoarthritis; UC-MSC Secretome; Randomized Controlled Trial; Sodium Hyaluronate; Intra-articular Injection
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: In this parallel assignment study, participants will be randomized to receive intra-articular injections of either UC-MSC-derived secretome or sodium hyaluronate.
Who Masked: Participant, Investigator
Masking Description: Participants and investigators will be blinded to treatment allocation. UC-MSC-derived secretome and sodium hyaluronate will be prepared and administered in a similar manner to ensure blinding is maintained during the study period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UC-MSC-Derived Secretome (Experimental): Participants receive intra-articular injection of UC-MSC-derived secretome
  Interventions: Drug: Sodium Hyaluronate (Hyalein)
- Sodium Hyaluronate (Active Comparator): Participants receive intra-articular injection of sodium hyaluronate
  Interventions: Biological: UC-MSC-Derived Secretome

INTERVENTIONS:
Biological: UC-MSC-Derived Secretome — Umbilical cord-derived mesenchymal stem cell secretome administered via intra-articular injection according to the study protocol.
  Arms: Sodium Hyaluronate
Drug: Sodium Hyaluronate (Hyalein) — Sodium hyaluronate administered via intra-articular injection as an active comparator.
  Other Names: Sodium Hyaluronate
  Arms: UC-MSC-Derived Secretome

SUMMARY:
This study is a randomized, double-blind, multicenter Phase II/III clinical trial designed to evaluate the effectiveness and safety of umbilical cord-derived mesenchymal stem cell (UC-MSC) secretome compared with sodium hyaluronate in patients with knee osteoarthritis. Knee osteoarthritis is a common degenerative joint disease that causes chronic pain and functional limitation. Participants will be randomly assigned to receive intra-articular injections of either UC-MSC-derived secretome or sodium hyaluronate. The study aims to assess improvements in knee pain, physical function, and overall clinical outcomes, as well as to evaluate the safety of the interventions over the study period.

DETAILED DESCRIPTION:
This multicenter, randomized, double-blind Phase II/III clinical study aims to compare the efficacy and safety of intra-articular UC-MSC-derived secretome with sodium hyaluronate in patients with Kellgren-Lawrence grade 2-3 knee osteoarthritis. Eligible participants will be randomly allocated to one of two treatment arms. Clinical outcomes will be evaluated using validated pain and functional assessment tools at predefined time points. Safety assessments will include monitoring of adverse events throughout the study period. The results of this study are expected to provide evidence regarding the potential role of UC-MSC-derived secretome as an alternative therapeutic option for knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with primary OA in one or both knees based on American College of Rheumatology (Clinical and Rheumatology criteria). If both knees have OA, the knee with the OA grade that falls within the inclusion criteria (grade 2-3) will be selected. If both knees meet the inclusion criteria, the knee with the highest grade and the one that is most uncomfortable will be chosen.
2. Males or females in the age range 40-70 years
3. Symptomatic knee OA (defined by pain at the affected joint for at least 3 months before inclusion and visual analog scale 40 - 70 mm on a 100 mm Visual Analog Scale (VAS).
4. Radiographic evidence of grade 2 to 3 osteoarthritis (OA) based on Kellgren and Lawrence radiographic criteria.
5. Body mass index between 18 - 30 kg/m2
6. Female participants of childbearing age who agreed to use accepted methods of contraception during the course of the study.
7. Ability to provide written informed consent and willing to participate the study

Exclusion Criteria:

1. Participants who, based on physical examination and clinical history (anamnesis), are in the active or acute phase of cardiac, pulmonary, hematological, hepatic, renal, systemic autoimmune, immunodeficiency, or coagulation disorders that may interfere with the administration of the study drug (Secretome or Sodium Hyaluronate) will be excluded,
2. Diagnosed with a meniscal rupture based on clinical history (anamnesis) and physical examination. If the anamnesis and physical examination show symptoms and signs of a meniscal rupture, further evaluation will be performed using ultrasound (USG),
3. Participants with significant axial deviation, defined by valgus or varus deformity observed during physical examination, will be excluded,
4. Participants with other pathological lesions on knee X-rays from the screening examination will also be excluded,
5. History of any form of secondary arthritis in the knee due to trauma,
6. History of surgery or major trauma to the knee joint
7. Has knee effusion,
8. Has any other inflammatory disorder of the knee joint
9. Diagnosed with active malignancy.
10. History of stem cell or secretome therapy.
11. Intra-articular injection of corticosteroid and/or prior treatment with Sodium Hyaluronate and/or platelet rich plasma (PRP) in past 3 months.
12. Use of NSAIDs and/or chondroprotective supplements, such as glucosamine and chondroitin sulfate, within 7 days before the trial, whether used orally, topically, or via injection,
13. Undergoing immunosuppressive therapy, or anticoagulant therapy, or corticosteroid therapy.
14. For women of child-bearing potential: positive pregnancy test or lactating (females who were planning pregnancy within the next year were excluded).
15. Enrolled in any other clinical trials within the past four weeks.
16. The principal investigator considers that the participant is ineligible for the clinical trial due to any reasons other than those listed above

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-16 (Estimated); Study Completion 2027-06-17 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in WOMAC Pain Subscale Score | Baseline to Week 24
  Change from baseline in knee pain assessed using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale.

SECONDARY OUTCOMES:
Change From Baseline in WOMAC Total Score | Baseline to Week 12
  Change from baseline in overall knee pain, stiffness, and physical function assessed using WOMAC total score.

CONTACTS AND LOCATIONS:
Overall Officials: Radiyati Umi Partan, MD, PhD, Study Chair — Universitas Sriwijaya
Locations (1):
- RSUP Dr. Mohammad Hoesin Palembang, Palembang, South Sumatera, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the primary and secondary outcome measures, including demographic characteristics, baseline clinical data, outcome scores, and adverse event data, will be shared. All data will be fully anonymized, with no direct identifiers, in accordance with applicable ethical and regulatory requirements.
Supporting Information: Study Protocol, SAP
Time Frame: De-identified individual participant data and supporting documents will be available beginning 6 months after publication of the primary study results and will remain available for up to 5 years.
Access Criteria: Access to de-identified IPD will be granted to qualified researchers who submit a methodologically sound research proposal. Requests will be reviewed by the study steering committee. Data will be shared under a data use agreement to ensure participant confidentiality and appropriate use of the data.
URL: https://rsmh.go.id